CLINICAL TRIAL: NCT05372926
Title: Evaluation of the Physiological Effects of High Flow Nasal Canulae Oxygen Therapy During Exercise in Patients With Fibrosing Interstitial Lung Diseases
Brief Title: Physiological Effects of HFNC During Exercise in Patients With Fibrosing Interstitial Lung Diseases
Acronym: HighFlowMusc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HighFlowMusc
Record Dates: First submitted 2022-04-06; First posted 2022-05-13 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Interstitial Lung Disease; Pulmonary Rehabilitation
Keywords: interstitial lung disease; nasal high flow oxygen therapy; endurance test; pulmonary rehabilitation
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: All patients were randomly allocated into two groups using the block randomization technique (blocks of eight patients) in a 1:1 ratio. In group A, a high-intensity constant work-rate endurance test using Venturi mask (VM) was performed on first, and a test using high-flow nasal canulae oxygen therapy (HFNC) was performed next. In group B, a high-intensity CWRET using HFNC was performed first, and a test using VM was performed next.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venturi mask (Experimental): Patients will be placed under oxygen therapy with Venturi mask at a constant flow of 15L/min and a set FiO2 of 50%. The real FiO2 will be mesured in the mask at rest.
  Interventions: Device: Ventury mask
- High flow nasal canulae (Experimental): Patients will be placed under high flow nasal canulae oxygen therapy with a constant flow of 50L/min and the real FiO2 provided by Venturi mask.
  Interventions: Device: high flow nasal canulae

INTERVENTIONS:
Device: high flow nasal canulae — high flow nasal canulae is a oxygen therapy technic which allows the administration of warmed and humidified oxygen with a flow up to 50L/Min and a monitored FiO2. Physiological previous studies reported various effects of this technic especially on work of breathing. In our study the investigators aim to test this physiological property during exercise.
  Arms: High flow nasal canulae
Device: Ventury mask — Ventury mask is a oxygen therapy technic which allows the administration with a mask of oxygen with a flow up to 15L/Min and a monitored FiO2.
  Arms: Venturi mask

SUMMARY:
in this study, the investigators aim to describe the effects of highflow nasal canulae oxygen therapy (HFNC) on respiratory muscle function during exercise in patients with fibrosing interstitial lung diseases (ILD) during an endurance test

ELIGIBILITY:
Inclusion Criteria:

* Cared for as part of a respiratory rehabilitation program (ADIR association)
* Presenting diffuse fibrosing interstitial pneumonitis, documented by CT scan data and whatever its etiology
* Presenting severe hypoxemia in ambient air (SpO2<90%) during an exercise test (6-minute walk test or functional exercise test)

Exclusion Criteria:

* Patient with a contraindication to carrying out a respiratory rehabilitation program
* Patient having presented an exacerbation of PID, pneumothorax or pneumomediastinum in the 3 months preceding potential inclusion
* Tracheostomized patient
* Patient with a contraindication to the placement of a nasogastric tube
* Pregnant or breastfeeding women or women of childbearing age without effective means of contraception (a pregnancy test will be carried out)
* Protected adult patient (guardianship or curatorship)
* Patient deprived of liberty by court or administrative decision
* Refusal of patient participation or consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-11-23 (Estimated); Study Completion 2024-11-23 (Estimated)

PRIMARY OUTCOMES:
Ptdi swing | during the intervention, at isotime
  To compare the change in transdiaphragmatic pressure between baseline and peak during inspiration (Ptdi swing) between HFNC and VM in patients with fibrosing Interstitial Lung Disease in stable state, at isotime.

SECONDARY OUTCOMES:
PTPdi | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of diaphragmatic pressure time product during a respiratory cycle (PTPdi)
PTPoeso | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of the respiratory "Pressure Time Product" during a respiratory cycle (PTPoeso)
Poeso swing | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of variation of oesophagal pressure between the base state and the peak (Poeso swing)
DeltaPtdi/DeltaEAdi | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of the electromechanical coupling of the diaphragm (ratio of variation of the transdiaphragmatic pressure by the variation of electrical activity of the diaphragm (EAdi) between the start of inspiration and the end of expiration, (DeltaPtdi/DeltaEAdi)
SmO2 | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of the measurement of tissue saturation in oxygen (SmO2) by "Near Infrared Spectrometry" (NIRS)
TcCO2 | during the intervention, at isotime
  on effort at isotime, comparison between HFNC and VM of transcutaneous CO2 measurement (TcCO2)
Tlim | during the intervention, at the end of endurance test
  Comparison of endurance time (Tlim) between HFNC and VM

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARTAUD-MACARI, MD, Principal Investigator — ADIR Association
Locations (1):
- ADIR association, Bois-Guillaume, France